CLINICAL TRIAL: NCT06358599
Title: The Impact of Neoadjuvant Chemotherapy on Survival Outcomes in Patients With Variant Histologies Who Underwent Radical Cystectomy: A Multicenter Study of the Turkish Urooncology Association
Brief Title: The Impact of Neoadjuvant Chemotherapy on Survival Outcomes in Patients With Variant Histologies Bladder Cancer Who Underwent Radical Cystectomy
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Cagri Akpinar, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: TUO-UR-21-01
Record Dates: First submitted 2024-03-13; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Bladder Cancer; Bladder Cancer Stage I; Bladder Cancer Stage II
Keywords: bladder cancer; variant histology; neoadjuvant therapy; radical cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant chemotherapy prior to radical cystectomy
  Interventions: Drug: Cisplatin
- radical cystectomy directly

INTERVENTIONS:
Drug: Cisplatin — Neoadjuvant cisplatin-containing combination chemotherapy was defined as the receipt of multiagent systemic chemotherapy initiated within 6 months prior to the date of radical cystectomy
  Other Names: neoadjuvant cisplatin containing combination chemotherapy
  Groups: Neoadjuvant chemotherapy prior to radical cystectomy

SUMMARY:
The World Health Organization 2016 bladder tumor classification reported that the diagnosis of variant histology has increased from 6% to 33% in the last 2 decades, and there is an increasing interest in investigating the effects on disease management, treatment options, and survival outcomes in bladder tumors with variant histology. In bladder tumors, variant histology is known to be more aggressive and has a worse prognosis than pure urothelial cancer, and most cases are muscle invasive at diagnosis. Neoadjuvant cisplatin-containing combination chemotherapy is known to improves overall survival in patients with urothelial cancers. However, it is unclear whether patients with non-pure urothelial cancer (variant) histology will also benefit from neoadjuvant chemotherapy. The investigators aimed to evaluate the role of Neoadjuvant cisplatin-containing combination chemotherapy in the final treatment plan and its impact on survival in patients with bladder cancer who were diagnosed with variant histology in the radical cystectomy specimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with squamous cell, micropapillary, nested variant, sarcomatoid, neuroendocrine, or plasmacytoid variant histology
* Patients who were non-metastatic at diagnosis
* Patients who completed staging and demographic data,
* Patients with pathological stage (p)T2 or high grade pT1, clinical stage (c)N0 or cN1, and underwent radical cystectomy

Exclusion Criteria:

* Although RC histopathology was variant histology, patients in whom variant histology was not detected in previously transurethral resection bladder pathology
* Patients who received therapies other than radical cystectomy (intravesical bacillus-calmette-guerin or chemotherapy) were excluded from the study.
* Patients with a concomitant diagnosis of upper urinary tract urothelial carcinoma
* Patients with histopathologically pure urothelial carcinoma

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: multiple tertiary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Change in survival outcomes at postoperative 2-year follow-up in patients with variant histology who received neoadjuvant chemotherapy before radical cystectomy. | 2 years from radical cystectomy surgery

SECONDARY OUTCOMES:
Factors associated with worse survival outcomes in cox-regression analysis at 2-year follow-up of all patients with variant histology who underwent radical cystectomy. | 2 years from radical cystectomy surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)